CLINICAL TRIAL: NCT06880107
Title: Genetic Variants of Annexin A2 and Cryptogenic Stroke
Acronym: GENANXVA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire, Amiens (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: PI2023_843_0150
Record Dates: First submitted 2025-03-11; First posted 2025-03-17 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Annexin A2; Stroke; Genetic Variants of Host; Fibrinolysis
Keywords: annexin A2; stroke; genetic variants; fibrinolysis
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- cryptogenic stroke (Experimental): cryptogenic stroke
  Interventions: Biological: blood withdrawal
- ischemic stroke (Experimental): ischemic stroke
  Interventions: Biological: blood withdrawal
- control subjects (Active Comparator): control subjects
  Interventions: Biological: blood withdrawal

INTERVENTIONS:
Biological: blood withdrawal — blood withdrawal

SUMMARY:
Stroke is the third most common cause of death in developed countries. Various mechanisms of ischemic stroke exist. However, in young population, in a third of cases, the cause of a stroke cannot be determined despite an extensive evaluation. Many studies have highlighted the link between stroke and fibrinolysis. Genetic variants of tPA and PAI-1 genes have been suggested to be the risk factors for stroke.

ANXA2 plays a pivotal role in plasmin generation and fibrinolysis. Several studies showed the role of ANXA2 and S100A10 subunits in regulation of fibrinolysis in vivo. Recently, the efficacy of recombinant ANXA2 for fibrinolytic therapy in a rat embolic stroke has been demonstrated. Some single nucleotide polymorphisms in ANXA2 gene could be associated with increased risk of stroke in sickle cell disease.

Therefore, these data invite us to test hypothesis that genetic variants of ANXA2 gene could be associated with ischemic stroke.

ELIGIBILITY:
Inclusion Criteria:

* Completed ischemic stroke defined as a rapidly developing focal neurologic deficit with no apparent cause other than a vascular origin that persisted beyond 24 hours in surviving patients
* Age from 18 years old

Exclusion Criteria:

* Transient ischemic attack
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2025-04-08 (Actual); Primary Completion 2027-04 (Estimated); Study Completion 2027-04 (Estimated)

PRIMARY OUTCOMES:
genetic variants of ANXA2 | day 1
genetic variants of S100A10 | day 1

SECONDARY OUTCOMES:
blood ANXA2 concentration | day 1
blood S100A10 concentration | day 1
concentration of Autoantibodies directed against ANXA2 | day 1
concentration of S100A10 directed against ANXA2 | day 1

CONTACTS AND LOCATIONS:
Locations (1):
- CHRU Amiens, Amiens, France

IPD SHARING:
Plan to Share IPD: No